CLINICAL TRIAL: NCT05294601
Title: Efecto de Los Juegos Infantiles de Alta Intensidad Comparado Con Los de Mediana Intensidad Sobre la regulación autonómica Cardiaca, Biomarcadores de Obesidad y composición Corporal en Niños y Niñas de 6 a 9 años Con Obesidad o Sobrepeso
Brief Title: Effect of High Intensity Children's Games Compared With Medium Intensityregulation, Obesity Biomarkers and Body Composition in Boys and Girls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Surcolombiana (Other)
Collaborators: Maciste Macias (Unknown); Gilberto Astaiza (Unknown)
Responsible Party: Principal Investigator, claudia rodriguez, Principal Investigator, Universidad Surcolombiana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3685
Record Dates: First submitted 2021-11-30; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Obesity, Childhood
Keywords: Obesity; children; High-Intensity Interval Training; Adipokines
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Three groups with nutritional interventions and recreational games and observation before and after of physiological variables needed in the outcomes.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIIG Group (Active Comparator): General nutritional recommendations will be suggested in an initial consultation with weekly telephone follow-up. The high intensity children's games program for 12 weeks, . In this group the activities will include 3 weekly sessions. . The games last 6 minutes with a 2 minute break, four games per session; which is the one established for children of these ages according to the cited authors. The session is divided into 5 minutes of warm-up, 36 minutes of intervention and 8 minutes of cool-down. The intensity varies between 85-95% of HR max. According to the equation of Tanka et., Al. HR max = 208-0.7 x age
  Interventions: Other: High-Intensity Interval Training
- MIIG Group (Active Comparator): : The interventions will be carried out by a graduate in physical education, recreation and / or sports and the main researcher. General nutritional recommendations will be suggested in an initial consultation with weekly telephone follow-up. The medium intensity physical activity program for 12 weeks (28). Medium intensity activities are very similar to those taught in physical education class. In this group the activities will include 3 weekly sessions, with six episodes of 10 min at 65% to 85% of maximum heart rate (HRmax) separated by 5 min of recovery.
  Interventions: Other: Medium-Intensity Interval Training
- Control Group (No Intervention): In this group, measurements will be made before, during and after the study. Neither medium nor high intensity interventions will be carried out in order to generate comparisons, control biases and confounding and interaction variables. However, the interventions that have been most beneficial in the intervention groups. It could be implemented in this study once the analysis between groups has been completed, according to the recommendations and follow-up by the ethics committee.

INTERVENTIONS:
Other: High-Intensity Interval Training — high intensity exercise with games
  Other Names: High Intensity Interval Games
  Arms: HIIG Group
Other: Medium-Intensity Interval Training — medium intensity exercise with games
  Other Names: Medium-Intensity Interval Games
  Arms: MIIG Group

SUMMARY:
To evaluate the effect of high intensity children's games compared with those of medium intensity on cardiac autonomic regulation, obesity biomarkers and body composition in Boys and Girls from 6 to 9 years old with Obesity or Overweight

DETAILED DESCRIPTION:
Childhood obesity presents as a multifactorial disease with serious health consequences . In the department of Huila, the situation with respect to cardiovascular diseases (CVD) and childhood obesity is similar to the whole country and is a public health problem, recognized by the territorial entities. Autonomic dysfunction associated with obesity has been documented in adults and has been related to eventual CVD. The evidence for autonomic dysfunction in children remains contradictory, as well as whether this eventual dysfunction can be reversed with training. High intensity interval training (HIIT) is considered efficient because it achieves similar benefits to moderate or low intensity aerobic exercise, but in less time in the adult population ; In children and adolescents, HIIT training strategies have been tested with excellent results, related to both body weight and cardiorespiratory fitness, and could improve autonomic control. In the case of children, HIIT must be transformed to adapt them to the corresponding age. Children's recreational games have a similar pattern to HIIT; with intervals of high intensity alternated by short periods of rest; However, high-intensity games take into account children's motor development and aim to achieve some benefits of HIIT without necessarily meeting its goals in terms of cardiovascular demand. The objective of this study is to evaluate the effect of high intensity children's games (HIIG) compared to medium intensity games (MIIG) on cardiac autonomic regulation and body composition in Boys and Girls from 6 to 9 years old with Obesity or Overweight from the city of Neiva-Huila.

In this research, an experimental type design, a randomized controlled clinical trial, will be applied. Reference population: Children between 6 and 9 years old with overweight and obesity, enrolled in educational institutions in Neiva. To determine the experimental sample, the inclusion and exclusion criteria will be applied. The participants will subsequently be randomly divided into two intervention groups and a control group. The sample for this study will be 35 children in the control group and 35 children in the HIIG group and 35 MIIG children, randomly chosen from among the boys and girls who have authorization from their tutors and who agree to participate voluntarily who have complied with the above criteria. The project will be developed in different four research phases: Phase I (Sensitization to parents and children), Phase II (Medical Assessment, Course navette test, Measurement of heart rate variability, Initial measurement of anthropometric parameters, body composition , salivary biomarkers for obesity), Phase III (high intensity children's games program will be for 12 weeks for the HIIG group and moderate intensity children's games program for the MIIG group according to Biljon et., al and Phase IV (Again, measurement of phase II variables.) It is hoped to determine if training through games changes cardiac autonomic control; inflammatory markers; as well as improve anthropometric variables and positively impact family lifestyles participants.

ELIGIBILITY:
Inclusion Criteria:

* Children from 6 to 9 years old with the consent of their parents or guardians and who agree to participate
* Clinically healthy verified by medical examination according to the Clinical Guide for cardiovascular evaluation prior to sports practice in pediatrics .
* Children with weight above the 85th percentile in relation to their growth and development scale for Colombia and as suggested by the study by Cole et., al
* Children who are included in the general social security system

Exclusion Criteria:

* Children with musculoskeletal diseases that limit or contraindicate physical activity.
* Children with chronic diseases (chronic asthma, kidney disease, diabetes), or who have received medications that alter body composition or in-sulin secretion such as glucocorticoids.
* Children who on medical examination have shown any history or evidence of heart disease
* Hypertension (defined as blood pressure above the 95th percentile for systolic or diastolic values)
* Diagnosed attention deficit hypersensitivity disorder
* Children who at the clinical discretion cannot participate or who have presented any symptoms (dyspnea, chest pain, palpitations, among others) during the physical fitness test.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-04-25 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
IL-6 salival levels | 12 weeks
  elisa test for IL-6 in saliva levels = 26.89 ± 9.97 pg/mL
TNF-α salival levels | 12 weeks
  elisa test for IL-6 in saliva levels= 43,56 ± 6,44 pg/mL
Leptin salival levels | 12 weeks
  ng / ml
Adiponectin salival levels | 12 weeks
  elisa test for Adiponectin (also known as Acrp30) is a hormone synthesized by white adipose tissue that mcg/ml participates in the metabolism of glucose and fatty acids. Salivary concentrations of 3.22-28.71 ng/ml
Insulin salival levels with elisa test | 12 weeks
  Hypoglycemic protein hormone that is secreted in the beta cells of the islets of Langerhans, the established reference ranges for adults are between 2.6 and 24.9μU/ml for insulin for adults, in children it is more variable and depends on age 0.20μU/ml and a maximum of 26.5μU/ml

SECONDARY OUTCOMES:
Heart rate variability | 12 weeks
  To assess the group-time effect of high-intensity games compared to medium-intensity games on heart rate variability in boys and girls aged 6 to 9 years with obesity or overweight.
fat mass percentage | 12 weeks
  Body composition: fat mass and muscle mass of boys and girls will be calculated based on the formulas of Slaughter et al. . and bioimpedance technique
Percentage of muscle mass | 12 weeks
  Body composition: fat mass and muscle mass of boys and girls will be calculated based on the formulas of Slaughter et al. . and bioimpedance technique

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Y Rodriguez-Triviño, Ph.D student, Principal Investigator — Universidad Surcolombiana-Universidad del Valle
Locations (1):
- Universidad Surcolombiana, Neiva, Huila Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Biljon A, McKune AJ, DuBose KD, Kolanisi U, Semple SJ. Short-Term High-Intensity Interval Training Is Superior to Moderate-Intensity Continuous Training in Improving Cardiac Autonomic Function in Children. Cardiology. 2018;141(1):1-8. doi: 10.1159/000492457. Epub 2018 Sep 18. PMID 30227396
- [Background] Aguilar Cordero MJ, Ortegon Pinero A, Baena Garcia L, Noack Segovia JP, Levet Hernandez MC, Sanchez Lopez AM. [REBOUND EFFECT OF INTERVENTION PROGRAMS TO REDUCE OVERWEIGHT AND OBESITY IN CHILDREN AND ADOLESCENTS; SYSTEMATIC REVIEW]. Nutr Hosp. 2015 Dec 1;32(6):2508-17. doi: 10.3305/nh.2015.32.6.10071. Spanish. PMID 26667697
- [Background] Garcia-Hermoso A, Cerrillo-Urbina AJ, Herrera-Valenzuela T, Cristi-Montero C, Saavedra JM, Martinez-Vizcaino V. Is high-intensity interval training more effective on improving cardiometabolic risk and aerobic capacity than other forms of exercise in overweight and obese youth? A meta-analysis. Obes Rev. 2016 Jun;17(6):531-40. doi: 10.1111/obr.12395. Epub 2016 Mar 7. PMID 26948135
- [Result] Amigo, T. R. R., & Labisa-Palmeira, A. (2020). Moderators of the effect of high-intensity and moderate-intensity games in school children on cardiorespiratory fitness and body composition. Motricidade, 16(2), 156-169.
- [Derived] Rodriguez-Trivino CY, Quintana S, Osorio-Velez CE, Garcia-Florez M. Effect of high-intensity childhood games on heart rate variability, saliva leptin concentrations, and body composition in children. Braz J Med Biol Res. 2025 Jun 16;58:e14479. doi: 10.1590/1414-431X2025e14479. eCollection 2025. PMID 40531756